CLINICAL TRIAL: NCT05682677
Title: Combined Neuromodulation and Cognitive Training for Post-mTBI Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Twamley, Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH-22-2-0045
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Depression; Mild Traumatic Brain Injury; Concussion, Brain
Keywords: brain stimulation; neuromodulation; transcranial magnetic stimulation; theta burst stimulation; TMS; TBS; rTMS; iTBS; cognitive training; cognitive rehabilitation
MeSH Terms: conditions — Depression; Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PACT+iTBS (Experimental): Personalized, Augmented Cognitive Training (PACT; 6 sessions over 4 weeks) + intermittent theta burst stimulation (iTBS; 20 sessions over 4 weeks)
  Interventions: Device: iTBS; Behavioral: Personalized, Augmented Cognitive Training (PACT)
- PACT+sham iTBS (Sham Comparator): Personalized, Augmented Cognitive Training (PACT; 6 sessions over 4 weeks) + sham intermittent theta burst stimulation (sham iTBS; 20 sessions over 4 weeks)
  Interventions: Device: sham iTBS; Behavioral: Personalized, Augmented Cognitive Training (PACT)

INTERVENTIONS:
Device: iTBS — iTBS over the left dorsolateral prefrontal cortex
  Arms: PACT+iTBS
Device: sham iTBS — sham iTBS over the left dorsolateral prefrontal cortex
  Arms: PACT+sham iTBS
Behavioral: Personalized, Augmented Cognitive Training (PACT) — 6 sessions of PACT

SUMMARY:
The primary goal of this clinical trial is to evaluate whether Personalized Augmented Cognitive Training (PACT) plus intermittent theta burst stimulation (iTBS) is effective for treating depression in Service Members, Veterans, and civilians who have sustained a mild TBI. Participants will receive PACT plus 20 sessions of iTBS or sham iTBS over 4 weeks. Assessments will occur at baseline, 2 weeks, 4 weeks, and 8 weeks. Researchers will compare the PACT+iTBS group to the PACT+sham iTBS group to see if PACT+iTBS is associated with more depression improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. All racial and ethnic groups
3. Ages 18 to 65
4. Military service members receiving treatment at NMCSD or civilians receiving treatment at UCSD Health
5. History of mild TBI (as defined by the DoD/VA criteria used in conjunction with the OSU TBI-ID method) over 3 months prior to study entry
6. Meets criteria for current Major Depressive Episode within the context of Major Depressive Disorder, per MINI
7. Score of 18 or higher on the HAMD-17, indicating moderate to severe depressive symptoms
8. Stable on psychiatric medications for 6 weeks, with no changes to psychiatric medications expected during the study period
9. No contraindications to TMS (passes the TMS Adult Safety Screening questionnaire)
10. No contraindications to MRI (passes MRI safety screening questionnaire)
11. Able to commit to the treatment schedule
12. Able to complete assessment procedures in English
13. Intact decision-making capacity and ability to provide voluntary informed consent

Exclusion Criteria:

1. History of moderate, severe, or penetrating TBI
2. History of other neurological condition unrelated to TBI, including but not limited to: conditions associated with increased intracranial pressure; space occupying brain lesions; cerebral aneurysm; stroke; transient ischemic attack within past two years; Parkinson's disease; Huntington's disease; dementia; multiple sclerosis; history of brain surgery; epilepsy; seizure except those therapeutically induced by electroconvulsive therapy (ECT) or a febrile seizure of infancy
3. Implanted medical devices including cardiac pacemaker, medication pump, aneurysm clip, shunt, stimulator, cochlear implant, electrodes, or any other metal object within or near the head (excluding the mouth) that cannot be safely removed
4. Active manic or psychotic illness per MINI
5. Current substance use disorder per MINI
6. Current active suicidal or homicidal ideation
7. Pregnant or intending to become pregnant within the study period; breastfeeding
8. Other sensory conditions or illnesses precluding participation in assessments or treatment
9. Current dose of lorazepam 2 mg or greater daily (or benzodiazepine equivalent) or any anticonvulsant due to the potential to limit iTBS efficacy
10. Taking medication that lowers seizure threshold
11. Previous failed treatment with rTMS, iTBS, or ECT
12. Completed >4 sessions of cognitive rehabilitation within the last 3 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | change over 8 weeks

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | change over 8 weeks
Neurobehavioral Symptom Inventory | change over 8 weeks
PTSD Checklist for DSM-5 | change over 8 weeks
Headache Impact Test | change over 8 weeks
Pittsburgh Sleep Quality Index | change over 8 weeks
WHO Disability Assessment Schedule | change over 8 weeks
Glasgow Outcome Scale - Extended | change over 8 weeks
PROMIS Cognitive Function Abilities Short Form | change over 8 weeks
Patient Global Impression of Change | rating at 8 weeks
  This measure asks the participant to rate their status since the start of the study from 1 (very much improved) to 7 (very much worse)
Traumatic Brain Injury Quality of Life | change over 8 weeks
  The Traumatic Brain Injury Quality of Life The Traumatic Brain Injury Quality of Life measurement system (TBI-QOL) is a TBI-specific extension of the NIH PROMIS and Neuro-QoL measures that includes 20 items measuring physical, emotional, social, and cognitive domains
D-KEFS Trail Making Test | change over 8 weeks
D-KEFS Color Word Interference Test | change over 8 weeks
WMS-IV Digit Span | change over 8 weeks
WAIS-IV Processing Speed | change over 8 weeks
Hopkins Verbal Learning Test - Revised | change over 8 weeks
UCSD Performance-Based Skills Assessment-Brief | change over 8 weeks
  The UCSD Performance-Based Skills Assessment-Brief is a performance-based measure that uses role play scenarios to assess capacity for financial and communication tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Twamley, PhD, Principal Investigator — UC San Diego
Locations (1):
- UCSD, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available via FITBIR.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following study completion; deidentified data available indefinitely.
Access Criteria: Via FITBIR request.
URL: https://fitbir.nih.gov